CLINICAL TRIAL: NCT04828083
Title: The Efficacy of Systemic Lidocaine Versus Ultrasound-guided Adductor Canal Block for Patients Undergoing Total Knee Arthroplasty: a Randomized, Double-blinded, Non-inferiority Study
Brief Title: Systemic Lidocaine Versus Ultrasound-guided Adductor Canal Block for Patients Undergoing Total Knee Arthroplasty
Acronym: ACBSL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1617319
Record Dates: First submitted 2021-03-08; First posted 2021-04-01 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Arthroplasty, Replacement, Knee; Total Knee Arthroplasty
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ultrasound-guided adductor canal block with local anesthetic (Active Comparator): Single shot Ultrasound-guided adductor canal block with 0.5% ropivacaine 30 ml
  Interventions: Drug: Saline IV
- Ultrasound-guided adductor canal block with saline (Sham Comparator): Single shot Ultrasound-guided adductor canal block with 30 mL of normal saline (Sodium chloride)
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — Intravenous lidocaine of 1.5 mg/kg bolus followed by a 1.5 mg/kg/h infusion continuing to the end of phase 1 of post anesthesia care unit
  Other Names: Lidocaine Hydrochloride
  Arms: Ultrasound-guided adductor canal block with saline
Drug: Saline IV — Intravenous saline of 1.5 mg/kg bolus followed by a 1.5 mg/kg/h infusion continuing to the end of phase 1 of post anesthesia care unit
  Other Names: Sodium chloride
  Arms: Ultrasound-guided adductor canal block with local anesthetic

SUMMARY:
The investigators are evaluating the postoperative outcomes in patients undergoing total knee arthroplasty that receive either systemic lidocaine or ultrasound-guided adductor canal block as part of their anesthetic plan.

DETAILED DESCRIPTION:
Patients scheduled to have total knee arthroplasty will typically receive a single shot adductor canal block to serve as the primary anesthetic and as part of a multi-modal post-operative analgesic plan. The use of adductor canal block is still limited to where trained anesthesiologists in regional anesthesia are available. There are other nonopioid analgesic adjuncts, such as Lidocaine, which is is widely available and is a very commonly used local anesthetic. A major advantage of lidocaine is that it is not associated with a significant side effect profile. Intravenous lidocaine which can be administered during surgery and/or after surgery has demonstrated anti-inflammatory effects and can significantly decrease the reliance on opioid use for adequate pain management in abdominal and spine surgeries. The addition of systemic lidocaine infusion as part of a multimodal analgesia strategy to minimize opioid related side effects might prove to be a useful combination for clinicians where adductor canal blocks are not a viable option. However, the level of evidence comparing the efficacy of intravenous lidocaine versus adductor canal block to reduce postoperative opioid consumption in patients undergoing TKA is limited. We hypothesized that there will be no meaningful clinical difference between systemic lidocaine and ultrasound-guided adductor canal block in the 24-hour postoperative analgesia period.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-3 patients undergoing primary, unilateral total knee arthroplasty

Exclusion Criteria:

* ASA PS classification of 4 or greater
* Pre-existing neuropathy
* Coagulopathy
* Chronic opioid consumption (>3 months)
* Infection at the site
* Known allergy to study medications (lidocaine)
* High grade atrioventricular block (cardiac conduction system impairment)
* A history of CVA/TIA
* Currently using lidocaine patches
* Known liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours
  Postoperative opioid consumption will be converted to equivalent dose of oral morphine.

SECONDARY OUTCOMES:
Pain Scores | up to 2 hours (post anesthesia recovery unit), 6 hours, 12 hours, and 24 hours after surgery.
  Patients were asked to rate their pain score during activity on a 11-point scale (0 = no pain to 10 = excruciating pain).
Quality of Recovery | 24 hours
  The QoR-15 questionnaire has 15 questions that assess patient-reported quality of a patient's postoperative recovery using a 11-point numerical rating scale that leads to a minimum score of 0 (poor recovery) and a maximum score of 150 (excellent recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Vendhan Ramanujam, M.D., Principal Investigator — Rhode Island Hospital, Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis GN, Rice DA, McNair PJ, Kluger M. Predictors of persistent pain after total knee arthroplasty: a systematic review and meta-analysis. Br J Anaesth. 2015 Apr;114(4):551-61. doi: 10.1093/bja/aeu441. Epub 2014 Dec 26. PMID 25542191
- [Background] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972
- See also: Intravenous lidocaine for acute pain: an evidence-based clinical update — https://doi.org/10.1093/bjaed/mkw008